CLINICAL TRIAL: NCT06257004
Title: Genome-wide Epistasis for Cardiovascular Severity in Marfan Study
Acronym: GEMS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Antwerp (Other)
Collaborators: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: 20/08/087; 1S81820N (Other Grant/Funding Number: FWO (Foundation for national research Belgium)); B3002021000292 (Other: Belgian number)
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-01

CONDITIONS: Marfan Syndrome; FBN1 Mutation
Keywords: p.Ile2585Thr;c.7754T>C; Rare disease; Aortopathies; TAAD; Congenital abnormalities; Genetic modifiers; Thoracic aortic disease; Thoracic aortic rupture
MeSH Terms: conditions — Marfan Syndrome; Rare Diseases; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. saliva collection (screening all subjects)
  2. bloodsampling (5% most extremes UMC and AMC participants)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AMC (Affected Mutation Carrier): FBN1 mutation (Marfan Syndrome) - Phenotype cardiovascular severe outcome
  Interventions: Genetic: Saliva collection (screening of all participants); Genetic: Bloodsampling
- UMC (Unaffected Mutation Carrier): FBN1 mutation (Marfan Syndrome) - Phenotype cardiovascular mild outcome
  Interventions: Genetic: Saliva collection (screening of all participants); Genetic: Bloodsampling

INTERVENTIONS:
Genetic: Saliva collection (screening of all participants) — All participants will give a salive sample (self-sampling kit) - selection of 25% extremes (UMC and AMC) participants for WGS and linkage analysis
Genetic: Bloodsampling — Based on the results of the WGS, a selection will be made of the 5% most extremes (UMC and AMC) participants for the iPSC-VSMC generation

SUMMARY:
Marfan syndrome (MFS) is an autosomal dominant connective tissue disorder with pleiotropic manifestations in the ocular, skeletal and cardiovascular systems. Morbidity and mortality are mostly determined by aortic root aneurysm dissection and rupture. Although mutations in FBN1, the gene coding for the extracellular matrix protein fibrillin-1, are the well-established genetic cause of this condition, there is a very poor correlation between the nature or location of the causal FBN1 mutation and the phenotypical outcome. Indeed, wide intra- and interfamilial phenotypical variability is observed. So, even with an identical primary mutation in all family members, the clinical spectrum varies widely, from completely asymptomatic to sudden death due to aortic dissection at a young age. The precise mechanisms underlying this variability remain largely elusive.

Consequently, a better understanding of the functional effects of the primary mutation is highly needed and the identification of genetic variation that modifies these effects is becoming increasingly important. In this project, we have carefully selected different innovative strategies to discover mother nature's own modifying capabilities with respect to Marfan syndrome aortopathy.

DETAILED DESCRIPTION:
In this project we will focus on the cardiovascular, or more specific, the TAAD (Thoracal Aorta Aneurysma Dissection) expressivity of the Marfan syndrome. The most frequent mutations in FBN1 (fibrilin-1 ), with significant aortopathy expressivity is p.Ile2585Thr; c.7754T>C and p.Ala882Val; c.2645C>T). We will limit the used population to p.Ile2585Thr; c.7754T>C mutation since this is the biggest population.

Marfan syndrome subjects carrying an identical FBN1 mutation show a variable aortopathy expressivity, even within one family. We hypothesize that the cardiovascular phenotypical variability is under control of genetic modifiers.

The first approach strategy involves ranking of carriers of the specific FBN1 mutation that present with significant variable aortopathy expressivity according to the severity of aortic aneurysma disease (based on Z-score, timing of surgery and manual expert curation). We will stratify these mutation carrying individuals in three groups: mild or no aortic disease (UMC, unaffected mutation carrier)), severely affected (AMC, affected mutation carrier), and participants with indeterminate data.

The second approach is the molecular characterisation of the 25% extreme cohort (AMC and UMC) using WGS (Whole Genome Sequencing) and linkage analysis.

Finally subjects peripheral blood mononuclear cells (PBMCs) of 10 severely affected mutation carrier (AMC) and 10 unaffected mutation carriers (UMC) as well as 2 controls will be reprogrammed to iPSCs (induced Pluripotential Stem Cells). These cells will finally be differentiated into VSMC's (VasculairSmoth Muscle Cells). The genomic integrity and identity of the iPSCs and the VSMCs will be validated using RT-PCR and immunocytochemistry.

Transcriptomic (i.e. RNA-sequencing) data will be acquired from these specific induced pluripotent stem cell-derived vascular smooth muscle cells (iPSC-VSMCs).

We will be able to filter the WGS data based on variant quality and location in genes that are differentially expressed when comparing the AMC and UMC iPSC-VSMCs, via the synchronization of both data types. This approach will allow us to identify the modifier gene. Once candidate modifier genes (and hence candidate modifier variants) have been identified, their modifying capacity will be functionally checked in relevant cell- or animal models. The choice of the model system will be determined based on the nature of the identified modifier. In an animal model, we will prove its effect by crossing an animal carrying the variant of interest with a MFS model, which should significantly alter the cardiovascular phenotype. Depending on the function and evolutionary conservation of the identified modifier gene, zebrafish or mouse models will be used.

Alternatively, the identified modifier will be functionally validated using the cutting-edge CRISPR/Cas9 genome editing technology in the available and thoroughly functionally characterized iPSC-VSMC lines.

Further evidence for a modifying role of the most interesting candidate genes will be obtained by performing targeted re-sequencing of these genes' coding and regulatory sequences in, again, the 25% most and least severely cardiovascular affected MFS cases of a large replication cohort consisting of more than 3000 clinically and molecularly (FBN1 mutation-positive) characterized index cases.

Whenever possible, segregation of the remaining candidate modifier variants with protection from TAAD will be investigated in available gDNA samples of the probands' relatives carrying the FBN1 mutation.

ELIGIBILITY:
Inclusion Criteria:

* Participants with proven mutation (p.Ile2585Thr;c.7754C>T) in the FBN1 gene

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: participants with Marfan syndrom
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-11-30 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Molecular characterization of the assembled 25% extreme ends cohort (UMC and AMC). | September 2023
  Whole Genome Sequencing (WGS) and linkage analysis will be used for this purpose

SECONDARY OUTCOMES:
Omics integration for modifier identification in the 5% extreme ends of the cohort (UMC and AMC) | September 2023
  The modifier genes will be identified by the generation of iPSC-VSMC's of MFS individuals from the 5% extreme ends of the spectrum.
Functional validation of the modifiers. | 2024
  For the validation of the modifiers the CRISP/Cas9 gene editing technology will be used.
Replication of the identified modifiers in a large MFS cohort Time frame: December 2024 | 2024
  The evidence for a modifying role of the most interesting candidate genes will be obtained by performing targeted re-sequencing of these genes again in the 25% most and least severely cardiovascular affected MFS cases of a large replication cohort consisting of more than 3000 clinically and molecularly characterized index participants.

CONTACTS AND LOCATIONS:
Overall Officials: Bart Loeys, Prof,MD,PhD, Principal Investigator — University Hospital, Antwerp; Paul Coucke, Prof,MD,Ing, Study Chair — University Hospital, Ghent
Locations (1):
- University Hospital Antwerp, Edegem, Prins Boudewijnlaan 43/6, Belgium

REFERENCES:
- [Background] Verstraeten A, Luyckx I, Loeys B. Aetiology and management of hereditary aortopathy. Nat Rev Cardiol. 2017 Apr;14(4):197-208. doi: 10.1038/nrcardio.2016.211. Epub 2017 Jan 19. PMID 28102232
- [Background] von Kodolitsch Y, De Backer J, Schuler H, Bannas P, Behzadi C, Bernhardt AM, Hillebrand M, Fuisting B, Sheikhzadeh S, Rybczynski M, Kolbel T, Puschel K, Blankenberg S, Robinson PN. Perspectives on the revised Ghent criteria for the diagnosis of Marfan syndrome. Appl Clin Genet. 2015 Jun 16;8:137-55. doi: 10.2147/TACG.S60472. eCollection 2015. PMID 26124674
- [Background] Groth KA, Gaustadnes M, Thorsen K, Ostergaard JR, Jensen UB, Gravholt CH, Andersen NH. Difficulties in diagnosing Marfan syndrome using current FBN1 databases. Genet Med. 2016 Jan;18(1):98-102. doi: 10.1038/gim.2015.32. Epub 2015 Mar 26. PMID 25812041
- [Background] Loeys BL, Dietz HC, Braverman AC, Callewaert BL, De Backer J, Devereux RB, Hilhorst-Hofstee Y, Jondeau G, Faivre L, Milewicz DM, Pyeritz RE, Sponseller PD, Wordsworth P, De Paepe AM. The revised Ghent nosology for the Marfan syndrome. J Med Genet. 2010 Jul;47(7):476-85. doi: 10.1136/jmg.2009.072785. PMID 20591885
- [Background] Braverman AC. Medical management of thoracic aortic aneurysm disease. J Thorac Cardiovasc Surg. 2013 Mar;145(3 Suppl):S2-6. doi: 10.1016/j.jtcvs.2012.11.062. Epub 2012 Dec 20. PMID 23260459
- [Background] De Backer J, Loeys B, Leroy B, Coucke P, Dietz H, De Paepe A. Utility of molecular analyses in the exploration of extreme intrafamilial variability in the Marfan syndrome. Clin Genet. 2007 Sep;72(3):188-98. doi: 10.1111/j.1399-0004.2007.00845.x. PMID 17718856
- [Background] Franken R, Teixido-Tura G, Brion M, Forteza A, Rodriguez-Palomares J, Gutierrez L, Garcia Dorado D, Pals G, Mulder BJ, Evangelista A. Relationship between fibrillin-1 genotype and severity of cardiovascular involvement in Marfan syndrome. Heart. 2017 Nov;103(22):1795-1799. doi: 10.1136/heartjnl-2016-310631. Epub 2017 May 3. PMID 28468757
- [Background] Renard M, Muino-Mosquera L, Manalo EC, Tufa S, Carlson EJ, Keene DR, De Backer J, Sakai LY. Sex, pregnancy and aortic disease in Marfan syndrome. PLoS One. 2017 Jul 14;12(7):e0181166. doi: 10.1371/journal.pone.0181166. eCollection 2017. PMID 28708846
- [Background] Granata A, Serrano F, Bernard WG, McNamara M, Low L, Sastry P, Sinha S. An iPSC-derived vascular model of Marfan syndrome identifies key mediators of smooth muscle cell death. Nat Genet. 2017 Jan;49(1):97-109. doi: 10.1038/ng.3723. Epub 2016 Nov 28. PMID 27893734